CLINICAL TRIAL: NCT00629733
Title: Clinical Trial to Evaluate the Tolerability and Pharmacokinetics of a New Ultra Low Molecular Weight Heparin (RO-14) Administered Subcutaneously Increasing Single-doses to Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rovi Pharmaceuticals Laboratories (Industry)
Responsible Party: Dr. Barbanoj, Hospital Santa Creu i Sant Pau
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ROV-RO14-2006-01
Record Dates: First submitted 2008-02-15; First posted 2008-03-06 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Healthy
Keywords: pharmacokinetics; ultra low molecular weight heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ro-14 (Experimental)
  Interventions: Drug: RO-14

INTERVENTIONS:
Drug: RO-14

SUMMARY:
Clinical trial to evaluate the tolerability and pharmacokinetics of a new ultra low molecular weight heparin (RO-14) administered subcutaneously increasing single-doses to healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers: male subjects aged between 18 and 45 years
2. Body weight: 65-75 Kg
3. Not meaningful abnormalities in physical examination and in clinical history
4. Without evidence of significant organic or psychiatric illness
5. Hemogram, biochemistry and coagulation in normal values established in the reference range of the local hospital laboratory
6. Vital signs (blood pressure, heart beat rate and body temperature) and EKG within normal range
7. Healthy volunteers who are not participating in another clinical trial or have not done so in the past 2 months
8. Not give blood in the last 4 weeks.
9. Healthy male volunteers who have not received heparin in the past
10. Healthy male volunteers who have accepted to participate in the study and have signed the written informed consent

Exclusion Criteria:

1. Previous history of alcoholism, drug dependency, drug abuse or habitual psychoactive drugs consumption
2. Important consumption of exciting drinks: alcohol consumption > 30 g/day; coffee, tea, cola > 5 /day
3. Allergy, idiosyncrasy or hypersensitivity to medicines
4. Healthy volunteers who are receiving another medication in the past 15 days
5. Positive serology of hepatitis B, C or HIV
6. Cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, hematologic, psychiatric, neurological and others events
7. Mayor Surgery in the last 6 months
8. Smoking > 10 cigarettes / day
9. Ethanol, cannabis, cocaine, amphetamine, benzodiazepine or opiate in urine
10. Healthy volunteers with a familiar history evident hemorrhagic episodes

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-12; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Main objective : To evaluate safety and tolerability of increasing single-doses to healthy male volunteers | safety parameters

SECONDARY OUTCOMES:
Secondary objectives : To evaluate pharmacokinetics profiles of each of single-doses. | anti-Xa activity

CONTACTS AND LOCATIONS:
Overall Officials: Dr Manuel Barbanoj, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital Santa Creu i Sant Pau, Barcelona, Spain